CLINICAL TRIAL: NCT06114511
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-M07D1 for Injection in Patients With HER2 Mutated, Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of BL-M07D1 in Patients With HER2-mutated, Locally Advanced or Metastatic Non-small-cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-201
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M07D1 (Experimental): Participants receive BL-M07D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion

SUMMARY:
This phase Ib/II study is designed to evaluate the safety, tolerability, pharmacokinetics, and efficacy of injectable BL-M07D1 in patients with HER2-mutated, locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol.
2. No gender limit.
3. Age: ≥18 years old and ≤75 years old.
4. expected survival time ≥3 months.
5. Histologically or cytologically confirmed, unresectable locally advanced or metastatic non-small cell lung cancer.
6. Confirmed known HER2-sensitive mutations, investigator-confirmed previous testing results, and trial site laboratory testing results were acceptable.
7. Patients in the advanced stage who had received platinum-based chemotherapy and immunotherapy concurrent or sequential therapy were unable to tolerate standard treatment or had disease progression during or after treatment.
8. Consent to provide archived tumor tissue or fresh tissue samples from primary or metastatic sites within 2 years for biomarker testing; Participants who were unable to provide tumor tissue samples could be enrolled if they met other inclusion and exclusion criteria after evaluation by investigators.
9. Must have at least one measurable lesion according to RECIST v1.1 definition.
10. ECOG score 0 or 1.
11. Toxicity of previous antineoplastic therapy has returned to grade 1 or less as defined by NCI-CTCAE v5.0 .
12. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%.
13. Organ function levels must meet the requirements.
14. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN.
15. Urine protein ≤2+ or ≤1000mg/24h.
16. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the start of treatment, serum/urine pregnancy must be negative, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Received chemotherapy, biological therapy, immunotherapy or other antitumor treatments within 4 weeks or 5 half-lives prior to the first dose (6 weeks for mitomycin and nitrosoureas; oral fluorouracil drugs, etc.).
2. Prior treatment with an ADC drug containing a camptothecin derivative (topoisomerase I inhibitor) as a toxin.
3. Presence of other gene mutations for targeted drug therapy.
4. A history of severe cardiovascular and cerebrovascular diseases.
5. Active autoimmune or inflammatory diseases.
6. Patients with other malignant tumors within 5 years before the first administration.
7. Unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening; Infusion-related thrombosis was excluded.
8. Patients with poorly controlled pericardial effusion, pleural effusion, peritoneal effusion, or pelvic effusion with clinical symptoms were judged by the investigator to be ineligible for enrollment.
9. Hypertension poorly controlled by antihypertensive drugs (systolic BP > 150 mmHg or diastolic blood pressure > 100 mmHg).
10. Current interstitial lung disease, drug-induced interstitial pneumonia, radiation pneumonitis requiring steroid therapy, or a history of these diseases.
11. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases). .
12. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any ingredient of BL-M07D1.
13. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
14. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > lower detection limit) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > lower detection limit).
15. Active infections requiring systemic therapy, such as severe pneumonia, bacteremia, sepsis, etc.
16. Had participated in another clinical trial within 4 weeks before the first dose (calculated from the time of the last dose).
17. Pregnant or lactating women.
18. Other circumstances considered by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M07D1.
Phase II: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-M07D1 to the first date of either disease progression or death, whichever occurs first.
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-M07D1 will be investigated.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-M07D1 will be investigated.
Ctrough | Up to 21 days after the first dose
  Ctrough is defined as the lowest serum concentration of BL-M07D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M07D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PHD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China